| Statistical | <b>Analysis Plan</b> |
|-------------|----------------------|
| Statistical | Allary Sis I lail |

AV005 Study Code

A Randomized, Double-blind, Single-Dose, 2-Period, Crossover Study to Assess the Efficacy of PT027 Compared with Placebo or Exercise-Induced Bronchoconstriction in Adult, and Advantage Subjects with Asthma (TYRF) Study to Assess the Efficacy of PT027 Compared with Placebo on In a in A ana (TYR)

Ana (TYR)

A

A Randomized, Double-blind, Single-Dose, 2-Period, Prossover Study to Assess the Efficacy of PT027 Compared with Placebo on Exercise-Induced Bronchoconstriction in Adult, and Adol Subjects with Asthma (TYREE)

This document must not be used to support any marketing author

A Randomized, Double-blind, Single-Dose, 2-Period, Crossover Study to Assess the Efficacy of PT027 Compared with Placebo on Exercise-Induced Bronchoconstriction in Adult and Andrew Subjects with Asthma (TVP Study to Assess the Efficacy of PT027 Compared with Placebo on

This document must not be used to support any marketing authoritization. 

3 of 45

Avillion

# Contents

| 1. | STUDY DETAILS | 9 | |
|---|---|---|---|
| 1.1 | Study objectives | 9 | |
| 1.1.1 | Primary objective | | |
| 1.1.2 | Secondary objective | 9 | |
| 1.1.3 | Safety objective | 9 | |
| 1.1.4 | Exploratory objective | 9 | |
| 1.2 | Study design | 9 | O<br>S |
| 1.3 | Number of subjects | 96 | |
| 1.3.1 | Randomization and stratification | 16 | |
| 1.3.2 | Sample Size Calculation | 16 | |
| 2. | ANALYSIS SETS | 17 | |
| ۷.<br>م | ANAL I SIS SETS | 17 | |
| 2.1 | Definition of analysis sets | I / | |
| 2.1.1 | All subjects enrolled. | I / | |
| 2.1.2 | All subjects randomized | 1 /<br>1 7 | |
| 2.1.3<br>2.1.4 | Sofoty analysis set | l /<br>17 | |
| 2.1. <del>4</del> | Safety analysis set | 1/ | |
| 2.2 | Protocol deviations | 18 | |
| 3. | DEMOGRAPHY AND SUBJECT CHARACTERISTICS VARIABLES | 18 | |
| 3.1 | Demographics | 18 | |
| 3.2 | Medical, asthma and smoking history. | 19 | |
| 3.3 | Concomitant medications | 19 | |
| 3.4 | Spirometry at study entry | 20 | |
| 3.5 | Treatment exposure | 20 | |
| 4. | Exploratory objective | 20 | |
| 4.1 | General Definitions Screening period | 20 | |
| 4.1.1 | Screening period . | 20 | |
| 4.1.2 | Crossover periods. | | |
| 4.1.3 | Relative time from exercise challenge test | 21 | |
| 4.1.4 | Relative time from first dose of randomized treatment | 21 | |
| 4.1.5 | Definition of baseline | 21 | |
| 4.1.6 | Absolute and percent change from baseline | | |
| 4.1.7 | Retreentage fall from post-dose pre-exercise baseline FEV <sub>1</sub> | | |
| 4.1.8 | Visit windowing | | |
| 4.1.9 | Imputation rules | | |
| 4.1.40 | Serial spirometry data | 24 | |
| <b>4</b> .2 | Primary Efficacy Measure | | |
| 4.2.1 | Maximum fall from post-dose, pre-exercise baseline in FEV <sub>1</sub> | | |
| 4.3 | Secondary Efficacy Measures | | |
| 4.3.1 | Derivation of responder status in post exercise FEV <sub>1</sub> (10% threshold) | 24 | |
| 4.4 | Exploratory Efficacy Measures. | 25 | |

| 4.4 | 4.1 Derivation of responder sta | atus in post exercise FEV1 (20% thresl | hold)25 |
|---|---|---|---|
| 4.4 | Time to recovery in post-e | xercise FEV <sub>1</sub> | 25 |
| 4.4 | Derivation of FEV <sub>1</sub> AUC <sub>0</sub> . | -30min | 26 |
| 4.5 | Safety variables | | 27 |
| 4.5 | 5.1 Vital signs | | 27 |
| 4.5 | 5.2 Adverse events (including | Serious Adverse Events) | 27 |
| 4.5 | | es | |
| 4.5 | 5.4 12-lead electrocardiogram. | | 31 |
| 4.0 | Other variables | | 31 |
| 4.0 | 6.1 Concomitant medications | | |
| 4.0 | 6.2 Withdrawal from study | | 31 |
| 4.0 | Screen Failures | | 32 |
| 4.0 | Maximum fall from post-d | lose, pre-exercise baseline in FEV <sub>1</sub> at V | Visit 232 |
| 5. | ANALYSIS METHODS | dpointde Characteristicsde Characteristicsde Characteristicsde characteristicsde characteristics | 33 × |
| 5.1 | Statistical Considerations | Jal. | 33 |
| 5.1 | 1.1 Estimands | <i>to.</i> | 33 |
| 5.1 | 1.2 Type I error control | ~ | 34 |
| 5.1 | 1.3 Treatment groups | | 34 |
| 5.2 | 2 Analysis methods | l all | 34 |
| 5.2 | 2.1 Subject Disposition | R div | 35 |
| 5.2 | 2.2 Demographic and Baseline | e Characteristics | 35 |
| 5.2 | 2.3 Treatment Exposure | | 36 |
| 5.2 | 2.4 Analysis of the primary en | dpoin();1 | 36 |
| 5.2 | 2.5 Analysis of the secondary | efficacy variables | 37 |
| 5.2 | 2.6 Analysis of safety variable | | 38 |
| 5.2 | 2.7 Analysis of exploratory va | riables | 39 |
| 5.2 | 2.8 Subgroup analysis | S <sub>II</sub> | 40 |
| 5.2 | 2.9 Supportive analysis | | 41 |
| 5.2 | 2.10 COVID-19 impacts | O O O O O O O O O O O O O O O O O O O | 41 |
| 6 | CHANGES OF ANALYS | IS FROM PROTOCOL | 44 |
| 6. | COVID-19 impacts | | 44 |
| 7 | DEFENE SEC | | |
| 7. | REFERENCES | | 45 |
| | eso. | | |
| | * De | | |
| | , 40° | | |
| | alst | | |
| × | | | |
| Mel | CHANGES OF ANALYS CHANGES OF ANALYS COVID-19 impacts REFERENCES REFERENCES | | |
| chi. | | | |
| 90. | | | |
| Khip. | | | |

## LIST OF TABLES

| | Table 1 Treatment sequences | .11 |
|---|---|---|
| | Table 2 Study Assessments and Procedures | .12 |
| | Table 3 Spirometry assessments relative to the maximal exercise test at Visit 1 | .14 |
| | Table 4 Spirometry assessments relative to the exercise challenge test and dosing at Visits 2, 3, and 4 | .15 |
| | Table 5 Laboratory Safety Variables | 30 |
| | Table 6 Subgroup Analysis | .40 |
| | of the state of th | |
| | LIST OF FIGURES | |
| | Figure 1: Study design | .10 |
| This doc | Table 2 Study Assessments and Procedures Table 3 Spirometry assessments relative to the maximal exercise test at Visit 1 | |

Statistical Analysis Plan Avillion

# LIST OF ABBREVIATIONS

| Abbreviation or special term | Explanation |
|---|---|
| AE | Adverse event |
| AUC <sub>0-30 minutes</sub> | Area under the curve from 0 to 30 minutes |
| BDA MDI (PT027) | Budesonide/albuterol metered-dose inhaler |
| BMI | Body mass index |
| ECG | Electrocardiogram |
| ECT | Body mass index Electrocardiogram Exercise challenge test Electronic case report form End-of-treatment |
| eCRF | Electronic case report form |
| EOT | End-of-treatment |
| | and a |
| FAS | Full Analysis Set |
| FEV <sub>1</sub> | Forced expiratory volume in 1 second |
| GINA | Full Analysis Set Forced expiratory volume in 1 second Global Initiative for Asthma International Conference on Warman Wattion |
| ICH | International Conference on Harmonization |
| ICS | International Conference on Harmonization Inhaled corticosteroid Investigational product Important protocol deviation Missing at random Metered-dose inhaler |
| IP | Investigational product |
| IPD | Important protocol deviation |
| MAR | Missing at random |
| MDI | Metered-dose inhaler |
| OAE | Other significant adverse event |
| PDV | Premature discontinuation visit |
| SABA | Short/rapid-acting β2-adrenoreceptor agonist |
| SAE & | Serious adverse events |
| SDTM | Study Data Tabulation Model |
| TC Used | Telephone contact |

| AMENDM |
|-------------|
| Date |
| AMENDM Date |

Statistical Analysis Plan Avillion

#### 1. **STUDY DETAILS**

### 1.1 **Study objectives**

### **Primary objective** 1.1.1

| Primary Objective: | Outcome Measure: |
|---|---|
| To assess the efficacy of a single dose of BDA MDI (160/180 μg) compared with placebo MDI on EIB in adult and adolescent subjects with asthma | The maximum percentage fall from post-dose, pre-exercise baseline in $FEV_1$ observed up to 60 minutes post-exercise challenge |

### **Secondary objective** 1.1.2

| Secondary Objectives: | Outcome Measures: |
|---|---|
| To further assess the efficacy of a single dose of BDA MDI compared with placebo MDI on EIB in adult and adolescent subjects with asthma | Percentage of subjects with a maximum percentage fall in $FEV_1$ post-exercise challenge of $<10\%$ |

#### 1.1.3 Safety objective

| Safety Objective: | Outcome Measures: |
|---|---|
| To evaluate the safety and tolerability of BDA MDI relative to placebo MDI on EIB in adult and adolescent subjects with asthma | Incidence of AEs/SAEs |

# 1.1.4

| adolescent subjects with asthma | |
|---|---|
| 1.1.4 Exploratory objective of the state of | |
| Exploratory Objective: | Outcome Measures: |
| To characterize the effect of BDAMDI 160/180 µg administered as a single-dose on bronchoconstriction compared with placebo | <ol> <li>Percentage of subjects with a maximum percentage fall in FEV<sub>1</sub> post-exercise challenge of &lt;20%</li> <li>Time to recovery, defined as the time from completion of the exercise challenge to the first measured post-exercise challenge FEV<sub>1</sub> value within 10% of the post-dose, pre-exercise challenge baseline FEV<sub>1</sub></li> <li>The percentage fall from baseline in FEV<sub>1</sub> at each time point within 60 minutes post-exercise challenge</li> <li>Post-exercise FEV<sub>1</sub> area under the curve from 0 to 30 minutes (AUC<sub>0-30min</sub>)</li> </ol> |

## 1.2 Study design

This is a multicenter, double-blind, randomized, placebo-controlled, 2-period, single-dose, crossover study. The study will consist of a screening period (Visit 1 and Visit 2) and 2

Statistical Analysis Plan Avillion

treatment visits (Visit 3 and Visit 4). A final follow-up visit will be conducted via a telephone call (TC) 3 to 5 days after the final in-clinic visit.

During the study, standardized exercise challenge tests (ECTs) are conducted according to American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines. At each visit, standard FEV<sub>1</sub> spirometry assessments will be performed relative to ECT and dosing, (before and after) as applicable. All spirometry and testing procedures are in accordance with current guidelines. A centralized spirometry data collection system incorporating a quality control program is used to reduce FEV<sub>1</sub> variability between and within subjects, and between study sites.

See Figure 1 for a graphical presentation of the study schema and Table 2 for a list of study assessments, and Table 3 and Table 4 for a list of the spirometry procedures conducted at the site, as per protocol.



Abbreviations: AE=adverse event; BDA=budesonide/albuterol; Conmeds=concomitant medication; EIB=exercise-induced bronchoconstriction; MDI=metered-dose inhaler; IP=investigational product; PDV=premature discontinuation visit.

Statistical Analysis Plan Avillion

Approximately 60 subjects will be randomized 1:1 to 1 of 2 treatment sequences (ie, A/B or B/A) as specified in Table 1 Treatment sequences

**Table 1 Treatment sequences** 

| | 1 abit 1 1 | i catificiti sequences | |
|---|---|---|---|
| | Treatment<br>sequence | Visit 3/Period 1 | Visit 4/Period 2 |
| | A/B | BDA MDI 160/180 μg (given as 2 actuations of BDA MDI 80/90 μg) | Placebo MDI (given as 2 actuations) |
| | B/A | Placebo MDI (given as 2 actuations) | BDA MDI 160/180 μg (given as 2 actuations of BDA MDI 80/90 μg) |
| This docum | Abbreviation | ns: BDA=budesonide/albuterol; MDI m BDA=budesonide/albuterol; MDI m REDA BLEDA BLE | Visit 4/Period 2 Placebo MDI (given as 2 actuations) BDA MDI 160/180 μg (given as 2 actuations of BDA MDI 80/90 μg) etered-dose inhaler. |
| | | THAL AND DRODDIETADY | 11 645 |

**Table 2 Study Assessments and Procedures** 

| | Screening <sup>a</sup> | | Double-blind Treatment Phase | | | Follow up |
|---|---|---|---|---|---|---|
| Visit | 1 | 2 | 3 | 4 | Unscheduled | |
| | I | 2 | Period 1 | Period 2 | Visit or PDV b (if | TC (3 to 5 days |
| Day | -14 to -8 <sup>a</sup> | -7 to -2 a | 1 | 8(±6) | Ø applicable) | after V4 or PDV |
| Informed consent/assent | X | | | ~ | | |
| Eligibility criteria | $X^c$ | X c | | ,iO' | | |
| Verify randomization criteria | | | $X^d$ | 100 | | |
| Routine clinical procedures | | | | 19, | | |
| Medical/surgical history | X | | | b | | |
| Demography | X | | | 1 0 | | |
| Alcohol consumption and smoking history | X | | | 0, | | |
| Physical examination | X | | . oʻ | X | X | |
| Height and BMI | X | | alle | | | |
| Weight | X | | 24 1100 | X | X | |
| Concomitant medications | X | X | 0, 20, | X | X | X |
| Routine safety measurements | | | | | | |
| Pregnancy test <sup>e</sup> | X | .(4) | ijo X | X | X | |
| Laboratory assessments f | X | | 10 | | | |
| Adverse events | X | X | X | X | X | X |
| Seated vital signs (blood pressure and heart rate) g | X | R Dauting | X | X | | |
| 12-lead ECG <sup>g, h</sup> | X | 10 | X | X | | |
| Efficacy measurements | | . Cill | | | | |
| Spirometry (FEV <sub>1</sub> ) <sup>g</sup> | X | X | X | X | | |
| Maximal exercise test h | $X^i$ | 10 | | | | |
| ECT with Treadmill h | | $X^{i,j}$ | $X^{i,j}$ | $X^{i,j}$ | | |
| Confirm FEV <sub>1</sub> stability <sup>k</sup> | . O | $X^k$ | $X^k$ | $X^k$ | | |
| Study treatment | of | | | | | |
| Randomization | .00 | | $X^d$ | | | |
| IP . | SUL | (placebo MDI) | X | X | | |

Abbreviations: β-hCG=beta-human chorionic gona@tropin; BMI=body mass index; ECG=Electrocardiogram; ECT=Exercise Challenge Test; EIB=exercise-induced bronchoconstriction; FEV1=Forced expiratory volume in 1 second; IP=Investigational Product; PDV=Premature discontinuation visit; TC=Telephone call; V=Visit.

Notes:

a The run-in periods at Screening are suggestions which can be shortened; the Screening and Double-blind Treatment Phase period must include at least 1 non-exercise test day between visit days.

<sup>&</sup>lt;sup>b</sup> Subjects who prematurely with thaw from the study will undergo a PDV.

Statistical Analysis Plan

\*\*Eligibility criteria: At V2 pre-dose FEV1 best value not exceeding ±20% of the best value measured at V1 pre-exercise; pre-exercise FEV1 ≥70% of preducted at V1 and V2; demonstration of EIB (at both V1 and V2). One retest will also be allowed for a lack of FEV1 drop (in pagative FIP extraore) at V1 and V2. demonstration of EIB (at both V1 and V2). One retest will also be allowed for a lack of FEV1 drop (ie, negative EIB outcome) at V1 only if the FEV1 drop is between 15% and <20%. Those subjects not meeting criteria will be considered screen failed.

d Subjects will be randomized at V3 to treatment if they demonstrate (at V3) a pre-exercise challenge  $FEV_1 \ge 70\%$  of predicted and a best pre-exercise challenge  $FEV_1$  that does not exceed  $\pm 20\%$  of the best pre-exercise challenge  $FEV_1$  at V1. that does not exceed  $\pm 20\%$  of the best pre-exercise challenge FEV<sub>1</sub> at V1.

e A serum pregnancy test (β-hCG) will be performed at V1, V4 and PDV; and a urine β-hCG test will be performed at V3 (for women of childbearing potential only). f Laboratory assessments (clinical chemistry, hematology and urinalysis).

g The spirometry (and related safety) assessments to be performed in association with the exercise challenge at V1 to V4 are described in detail in Table 3 and Table 4 for details.

h Heart rate to be monitored continuously during the exercise challenge and until 60 minutes after completion.

After V1. every attempt should be made to have subsequent ECTs started ±2 hours of the timing of the maximal exercise text done at V1.

<sup>j</sup> At V2, V3, and V4, an ECT will be conducted 30 ( $\pm$ 5) minutes after IP administration.

\* After VI, every attempt should be made to have subsequent ECTs started ±2 hours of the timing of the maximal exercise telePalone at VI.

\* At V2, V3, and V4, an ECT will be conducted 30 (±5) minutes after IP administration.

\* The pre-dose, pre-exercise challenge best FEV; value measured at each denoted visit (performed before exercise gladlenge) should not exceed ±20% of the pre-dose, pre-exercise challenge best FEV; value measured at VI.

\*\*EXECUTE: A provided in the pre-dose of the pre-dose of the pre-dose, pre-exercise challenge best FEV; value measured at VI.

\*\*EXECUTE: A provided in the pre-dose of the pre-dose, pre-exercise challenge best FEV; value measured at VI.

\*\*EXECUTE: A provided in the pre-dose of the pre-dose, pre-exercise challenge best FEV; value measured at VI.

\*\*EXECUTE: A provided in the pre-dose, pre-exercise challenge best FEV; value measured at VI.

\*\*EXECUTE: A provided in the pre-dose, pre-exercise challenge best FEV; value measured at VI.

\*\*EXECUTE: A provided in the pre-dose, pre-exercise challenge best FEV; value measured at each denoted visit (performed before exercise challenge) should not exceed ±20% of the pre-dose, pre-exercise challenge best FEV; value measured at each denoted visit (performed before exercise challenge) should not exceed ±20% of the pre-dose, pre-exercise challenge best FEV; value measured at each denoted visit (performed before exercise challenge) should not exceed ±20% of the pre-dose, pre-exercise challenge best FEV; value measured at each denoted visit (performed before exercise challenge) should not exceed ±20% of the pre-dose, pre-exercise challenge best FEV; value measured at each denoted visit (performed before exercise challenge) should not exceed ±20% of the pre-dose, pre-exercise challenge best FEV; value measured at VI.

\*\*EXECUTE: A provided in the pre-dose, pre-do

Table 3 Spirometry assessments relative to the maximal exercise test at Visit 1

| | Pre-e | exercise chal | lenge | Maximal exercise test | Post-exercise challenge | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time (minutes) | -50 | -35 (±5) | -5 (±3) | 0 | 5 (±3) | 10 | 15 | 20 | 30 | 40 | 45 | 60 |
| Assessments | (±15) | | | | | (±3) | (€3) | (±5) | (±5) | (±5) | (±5) | (±5) |
| Seated vital signs (BP and HR) | $X^{a}$ | | | | | | | X | | X | | $X^{b}$ |
| 12-lead ECG | $X^c$ | | | | | 787 | | | | | X | |
| Spirometry <sup>d</sup> | | X | X | | $X_{\bullet}$ | X | X | | X | | | X |
| Exercise challenge <sup>e</sup> | | | | X | 00 | | | | | | | |
| $HR$ monitoring $^f$ | | | | X | | | | | | | | X |
| Concomitant medication monitoring | X | | | | | | | | | | | X |
| AE monitoring | X | | | | | | | | | | | X |

Abbreviations: ACQ-7=Asthma Control Questionnaire 7, AQLQ+12= Asthma Quality of Life Questionnaire for 12 years and older; ECG=electrocardiogram; FEV1= forced expiratory volume in 1 second; IP=investigational product; min=minute; PAQLO=Pediatric Asthma Quality of Life Questionnaire

a. Notes:

b. a Vital signs should be recorded with the subject in the seated position and after 10 minutes of rest.

b Seated vital signs at the 60-minutes post-exercise challenge time point should be recorded 5-10 minutes AFTER the last PFT (ie, 65 minutes [±5 minutes]).

<sup>&</sup>lt;sup>c</sup> 12-lead ECG recording at the pre-exercise challenge time point should be conducted after 10 minutes of rest.

d Every attempt should be made to perform the first pre-exercise (and pre-dose at Visits 2 to 4) spirometry measurement prior to 11:00 AM consistently across Visits 1 through 4 visit (ie,  $\pm 1$  hour of the timing of the initial assessment at Visit 1).

<sup>&</sup>lt;sup>e</sup> After Visit 1, every attempt should be made to have the subsequent ECTs done  $\pm 2$  hours of the timing of the maximal exercise test done at Visit 1.

g. f Heart rate will be monitored continuously during the maximal exercise test and intermittently after maximal exercise test until 60 minutes after completion of the exercise challenge (ie, intermittently during PFTs).

Table 4 Spirometry assessments relative to the exercise challenge test and dosing at Visits 2, 3, and 4

| | Pre-dose Dose Post-dose Post-exercise challenge | | | | | ıge | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time (minutes) | -50 | -5 (±3) | 0 | 30 | ECT | 5 (±3) | 10 | 15 | 20 | 30 | 40 | 45 | 60 |
| Assessments | (±15) | | | (±5) | | | (±3) | (±3) | (±5) | (±5) | (±5) | (±5) | (±5) |
| Seated vital signs (BP and HR) | $X^{a}$ | | | | | | | | OX | | X | | $X^{b}$ |
| 12-lead ECG | $X^{c}$ | | | | | | | ijo | | | | X | |
| Spirometry <sup>d, e</sup> | | $X^{d, e}$ | | X | | X | X | OX | | X | | | X |
| Administer study drug <sup>f</sup> | | | X | | | | Kno | , | | | | | |
| Exercise challenge <sup>g</sup> | | | | | X | | ot | | | | | | |
| HR monitoring <sup>h</sup> | | | | | X | ioi | | | | | | | X |
| Concomitant medication monitoring | X | | | | 87 | 311Co | | | | | | | X |
| AE monitoring | X | | | | 7 86 | | | | | | | | X |

Abbreviations: AE=adverse event; BP=blood pressure; ECG=electrocardiogram ECF exercise challenge test; HR=heart rate; PFT=pulmonary function test.

Notes:

Notes:

a Vital signs should be recorded with the subject in the seated position and after 10 minutes of rest.

c 12-lead ECG recording at pre-dose time point should be conducted after 10 minutes of rest.

<sup>&</sup>lt;sup>b</sup> Seated vital signs at the 60-minutes post-exercise challenge time point should be recorded 5-10 minutes AFTER the last PFT (ie, 65 minutes [±5 minutes]).

<sup>&</sup>lt;sup>d</sup> At Visits 2 through 4, if the FEV<sub>1</sub> criteria are not met in the first spirometry measurement (ie, 5 minutes pre-dose), 1 optional pre-dose spirometry measurement can be repeated after 30 minutes of the initial attempt. If first pre-dose  $FEV_1$  fulfill all criteria, then the subject can proceed to dosing.

<sup>&</sup>lt;sup>e</sup> Every attempt should be made to perform the first pre-exercise spirometry measurement prior to 11:00 AM consistently across Visits 1 through 4 visit (ie,  $\pm 1$ hour of the timing of the initial spirometry performed at Visit 1).

f At Visit 2, subjects will receive placebo; while at Visit 3 and Visit 4 they will receive IP (BDA MDI or placebo MDI) depending on their randomization assignment.

g After Visit 1, every attempt should be made to have the subsequent ECTs done  $\pm 2$  hours of the timing of the maximal exercise test done at Visit 1.

h Heart rate will be monitored continuous during the ECT and intermittently after ECT until 60 minutes after completion of the exercise challenge (ie, intermittently during PFTs).

### 1.3 Number of subjects

The target population will be outpatient subjects 12 to 70 years of age with asthma and exercise-induced bronchoconstriction (EIB).

#### 1.3.1 Randomization and stratification

At Visit 3, eligible subjects are randomized (1:1) to receive 1 of 2 treatment sequences (BDA MDI 160/180 / Placebo MDI or Placebo MDI / BDA MDI 160/180). Randomization is centralized and stratified by age (adults: 18 years to 70 years; adolescents: 12 years to 17 years) and background ICS therapy (ICS or non-ICS).

Two subgroups of approximately equal size are included in the study, one subgroup of subjects currently treated with short/rapid-acting β2-adrenoreceptor agonist (SABA) prn alone, and a second subgroup on low-to-medium-dose inhaled corticosteroid (ICS) maintenance therapy (according to Global Initiative for Asthma [GINA] guidelines) and SABA prn.

1.3.2 Sample Size Calculation

Prior studies of a similar design have randomized subjects who experience exercise-induced

symptoms without other generalized asthma symptoms. Other studies have permitted enrollment of those subjects experiencing exercise symptoms who may or may not be subjects with asthma (Bonini et al 2013). This study will only randomize subjects with asthma who are receiving background therapy for asthma (SABA prn alone; low-to-medium dose ICS plus SABA prn). Sub-analyses will be conducted on the primary endpoint for each of these subgroups of equal size.

Power calculations are based on the properties of the primary endpoint, the maximum

percentage fall from post-dose, pre-exercise baseline in FEV<sub>1</sub> observed up to 60 minutes postexercise challenge. A sample size of 30 subjects in each subgroup will provide a 92% probability to detect a difference of -9% between BDA MDI versus placebo MDI, within each of the 2 subgroups of interest (SABA prn alone; low-to-medium dose ICS plus SABA prn), assuming 2-stded, 5% level tests and a within-subject standard deviation of 10%. Randomization of 60 subjects in total will provide >99% overall probability to detect a difference of -9% between BDA MDI versus placebo MDI assuming a 2-sided, 5% level test and an estimated within-subject standard deviation of 10%. Since all subjects randomized in the study will be receiving background therapy for asthma, a more conservative estimate of variability and treatment effect has been assumed compared to studies of similar design (Ostrom et al 2015).

#### 2. ANALYSIS SETS

#### 2.1 **Definition of analysis sets**

#### 2.1.1 All subjects enrolled

tension of such application The all enrolled subject population includes patients who have provided signed informed consent for the study. The enrolled population will be used to present overall descriptive summaries of subject disposition.

#### 2.1.2 All subjects randomized

The all subjects randomized population includes all subjects who have been randomized in the trial, irrespective of having at least 1 primary efficacy assessment (see 2.1.3). This population will be used to describe subject allocation and exclusion from the full and safety analysis sets, and stratification factors at randomization. Descriptive summaries based on the randomized population will be grouped by randomized treatment sequence.

population will be grouped by randomized treatment sequence.

2.1.3 Full analysis set

The full analysis set (FAS) is defined as all subjects who are randomized to treatment and have the following available measurements at either Vicit 3 or Visit 4:

- Pre-dose baseline FEV<sub>1</sub>
- Post-dose, pre-exercise baseline FEV<sub>1</sub>

Please see section 4.1.5 for the definitions of baseline FEV<sub>1</sub>. Subjects will be analyzed according to the treatment they were assigned as per the randomization scheme regardless of the actual IP received.

Additionally, data suspected to be fraudulent will be reviewed on a case-by-case basis and may lead to exclusion from the FAS. Such exclusions will be fully documented and all data will be readily available in the SDTM and ADaM datasets.

All effector analyses will be conducted on the FAS.

## Safety analysis set

The safety analysis set is defined as all subjects receiving any amount of the IP. Subjects will be classified on the basis of treatment they actually received within each treatment period regardless of the treatment they were randomized to. Occurrences of safety events will be


summarized under the actual treatment corresponding to the treatment period of which the event occurred. Further details on treatment assignment for occurrence safety data is described in Section 5.2.6.

tension of such application All safety summaries will be based on the safety analysis set. Additionally, data suspected to be fraudulent will be reviewed on a case-by-case basis and may lead to exclusion from the safety analysis set. Such exclusions will be fully documented and all data will be readily available in the SDTM and ADaM datasets.

#### 2.2 Protocol deviations

Important protocol deviations (IPDs) are defined as a subset of protocol deviations that may significantly affect the completeness, accuracy, and/or reliability of the study data or that may significantly affect a subject's rights, safety, or well-being. All protocol deviations classified as important will be listed along with the full deviation term and coded form as provided in the SDTM data. The important deviations will be summarized in terms of the number and percentage of subjects meeting the pre-defined protocol deviation coded. IPDs will be identified by the sponsor prior to the primary database lock and unblinding of the study results.

A per protocol analysis excluding subjects with important protocol deviations is not planned. However, any subjects or site activity identified or suspected to be fraudulent (e.g. subjects who are enrolled on this clinical study more than once or another interventional clinical study, subjects re-enrolling onto the study or fabricated data) will be excluded from the analysis populations defined in section 2.1. Such instances will be reviewed on a case-by-case basis and fully documented by the Sponsor prior to unblinding.

All subjects who failed any inclusion/exclusion criteria will be listed along with details of the failed criteria. This information will also be summarized in terms of the number and percentage of subjects falling any of the inclusion/exclusion criteria and will be based on the FAS.

Any miss-stratified subjects will be identified as important protocol deviations. All subjects who are randomized and are part of the FAS will be analyzed according to the strata they were allocated to in IVRS/IWRS, as opposed to their actual strata.

# **Demography and Subject Characteristics Variables**

# **Demographics**

The following demographic characteristics are collected at Visit 1.

Ethnicity\*

- Race\*
- Sex

on such application of such application lo Additionally, age is collected at randomization. The age group strata will be derived based on the age at randomization and will be categorized as

Adolescents:  $\geq 12$  to 17 years

Adults: ≥ 18 years

Subjects must meet the eligibility criteria, assessed during screening, to be randomized to treatment. The list of inclusion and exclusion criteria are provided in the protocol. Eligibility criteria not met are collected on the eCRF.

Vital signs collected at Visit 1 includes height (cm), weight (kg) and a derivation of body mass index (BMI) (kg/m<sup>2</sup>), as collected in the eCRF

# Medical, asthma and smoking history 3.2

Medical (including surgical), asthma and smoking history are recorded on the eCRF at Visit 1. General medical history will be categorized into past and current medical history. Current medical history will be defined as a condition that is either classified as on-going, or ending after the first dose of randomized treatment.

Additionally, the time since diagnosis of asthma (years) will be calculated as

(Date of first dose of randomized treatment (Visit 3) - Date of diagnosis of

Partial dates for the above calculations will be handled as per section 4.1.9.

# **Concomitant medications**

Albeoncomitant medication will be recorded on the eCRF throughout the study. Disallowed medications will be identified by a physician or Avillion medical director (or designee) on review of the data which will be completed prior to database lock. All identified medications which are disallowed will be considered for flagging as an IPD during the protocol deviation reviews, prior to database lock and unblinding.


<sup>\*</sup> Race and/or ethnicity will be collected depending on local regulations.

### 3.4 Spirometry at study entry

Lung function measurements of FEV<sub>1</sub> (L), FVC (L), FEV<sub>1</sub>/FVC (%) are recorded at screening Jaments for Jaments can be rescheduled if the mosessments can be rescheduled if the mosessments can be rescheduled if the mosessments can be retested an upper mirection.

If any of the spirometry criteria are not met at Visit 1, subjects can be retested within 2 to 10 days of the initial visit. Only 1 retest will be permitted for reasons related to technical ison (ie, acceptability) and/or pre-exercise FEV₁ ≥70% predicted, prior \*\*

3.5 Treatment are

Treatment exposure

Treatment exposure and dosing information is collected on the eCRF. The time of IP administration occurring at the scheduled visits will be collected in the

### PRIMARY AND SECONDARY VARIABLÉS 4.

#### **General Definitions** 4.1

#### Screening period 4.1.1

Screening assessments are collected at Visit 2 and Visit 2 (see Table 2). One retest is allowed for a lack of FEV1 drop (ie, negative EIR outcome) at V1, these retests are defined as Visit 1a in the raw data.

Lung function data collected at Visit la should be used to represent the Visit 1 value for subjects in descriptive summaries at screening.

## 4.1.2 Crossover periods

Patients will be randomized to a particular sequence and will receive the first treatment in their sequence at Visit 3 and second treatment at Visit 4. Period 1 corresponds to the results collected at Visit and Period 2 corresponds to results collected at Visit 4. Patient data will be grouped by the treatment they received in each period in the study outputs. The below table represents planned treatment group assignment based on randomized sequence and crossover

| Randomized Treatment Sequence | Planned treatment group | |
|---|---|---|
| • | Period 1 (Visit 3) | Period 2 (Visit 4) |
| BDA MDI 160/180 /<br>Placebo MDI | BDA MDI 160/180 | Placebo MDI |

| Placebo MDI / | Placebo MDI | BDA MDI 160/180/ |
|-----------------|-------------|------------------|
| BDA MDI 160/180 | | |

device at site. The start and stop Times of spirometry assessments are collected in the times of the exercise challenge test are collected in the eCRF.

#### 4.1.4 Relative time from first dose of randomized treatment

In order to calculate the baseline FEV<sub>1</sub> endpoints (4.1.5), the time relative to first dose of randomized treatment, within the specific visit (visit 3 and 4) will be calculated as:

[Relative time from first dose (minutes)] = [time of assessment (HH:mm)] – [time of first dose (HH:mm)].

The relative time from first dose of placebo will be calculated at Visit 2 and will use the same derivation provided above.

Times of spirometry assessments and times of dosing at the scheduled visits will be collected in the device at site.

### Definition of baseline 4.1.5

## Period specific post-dose pre-exercise baseline 4.1.5.1

Post-dose pre-exercise baseline is defined as the FEV<sub>1</sub> result taken post-dose of randomized treatment and prior to the exercise challenge test conducted at Visit 3 and Visit 4 (approximately occurring 30 minutes post dose of IP, Table 4). The post-dose pre-exercise baseline is period specific and therefore will be calculated at each Visit 3 and Visit 4.

The post-dose pre-exercise baseline will be used to calculate the primary, secondary and

Only lung function measures Only lung function measurements of acceptable, or borderline acceptable quality will be considered for the assignment of baseline. If all post-dose pre-exercise spirometry efforts available are of an unacceptable quality, then the baseline will be missing.

#### 4.1.5.2 Period specific pre-dose baseline

The period specific pre-dose baseline is defined as the spirometry measurement taken prior to dosing of randomized treatment, which should occur at 5 minutes pre-dose of IP (Table 4). The period specific pre-dose baseline will be calculated separately at Visit 3 and Visit 4.

of such application The period specific pre-dose baseline will be included as a covariate in parametric analyses of the primary, secondary and exploratory endpoints.

Only lung function measurements of acceptable, or borderline acceptable quality should be considered for the assignment of baseline. If all pre-dose spirometry efforts available are of an unacceptable quality, then the baseline will be missing.

The period specific pre-dose baseline will additionally be used to calculate changes from baseline in safety endpoints of vital sign parameters and ECG parameters.

#### 4.1.5.3 Average pre-dose baseline

The average pre-dose baseline will be calculated as the average of the non-missing period specific pre-dose baseline result for each subject. The average pre-dose baseline will be included as a covariate in parametric analyses of the primary, secondary and exploratory endpoints.

# Absolute and percent change from baseline 4.1.6

Absolute change from baseline outcome variables is computed as

Absolute change from baseline (post-baseline value – baseline value).

Percent change from baseline is computed as

Percentage change from baseline =  $\lceil (post-baseline \ value - baseline \ value) / baseline$ 

If either the post-baseline value or the baseline value is missing, then the absolute/percent change from baseline value will also be set to missing. Unacceptable quality spirometry measurements will not be used in the calculation of absolute/percentage change from baseline.

# Percentage fall from post-dose pre-exercise baseline FEV<sub>1</sub>

Percentage fall from post-dose pre-exercise baseline FEV<sub>1</sub> will be used to calculate primary, secondary and exploratory lung function endpoints and is defined as

[Percentage fall from post-dose pre-exercise baseline] = [(post-dose pre-exercise baseline value – post-exercise value) / post-dose pre-exercise baseline value] × 100%.

The percentage fall from post-dose pre-exercise FEV<sub>1</sub> will be calculated at each post-exercise timepoint at Visits 2, 3 and 4.

sion of such application If either the post-baseline value or the baseline value is missing, then the percentage fall from baseline value will also be set to missing. Unacceptable quality spirometry measurements will not be used in the calculation of percentage fall from baseline.

#### 4.1.8 Visit windowing

Due to the design of this trial, there will be no visit windowing applied other than the identification of baseline as per definitions given in section 4.1.5. Any unscheduled visits which may occur will not be used in analyses, however all data will be listed where appropriate.

### 4.1.9 **Imputation rules**

When determining whether concomitant medication or adverse event emergence is pre- or post-randomized treatment, the following imputation methods will be applied.

## Partial end date

- 1. If missing day [--/mm/yyyy] then impute as minimum (the end of the month, end of study participation}.

  2. If missing month [--/--/yyyy] then impute as minimum {[31/12/yyyy], end of study
- participation}
- 3. If completely missing, then set to end of study participation.

## Partial start date

- 4. If missing day [--/mm/yyyy] then impute as the minimum of:
  - If mm/yovy is the same as the dose date of BDA MDI then set to dose date of BDAMDI; else if mm/yyyy is the same as the dose date of post-randomization Riacebo MDI then set to dose date of Placebo MDI; else set to 01/mm/yyyy
  - End date of medication/ event (after partial date handling has been applied).
- 5. If missing month [--/--/yyyy] then impute as the minimum of:
  - If yyyy same year as BDA MDI then set to date of BDA MDI dose; else if yyyy same year as post-randomization Placebo MDI dose date set to dose date of Placebo MDI; Else set to start of the year [01/01/yyyy].
  - End date of medication/ event (after partial date handling has been applied).
- 6. If completely missing, then impute as the minimum of:
  - Date of first dose of BDA MDI, unless missing then date of first dose of randomized Placebo MDI.
  - End date of medication/ event (after partial date handling has been applied).

This imputation method is defined to enable the classification of adverse events and concomitant medications as pre- or post-treatment for reporting in summary tables. The above imputation process will additionally assign the occurrence to the BDA MDI treatment group, unless it can be unequivocally determined otherwise, based on the partial information collected. The raw, original dates will be presented in any listings produced.

The primary endpoint of maximum percentage fall from post-dose, pre-exercise baseline in FEV<sub>1</sub> observed up to 60 minutes post-exercise challenge will have missing values imputed as part of a sensitivity analysis. Please refer to Section 5.2.9 for further details on this imputation

Serial spirometry data collected by the device will be conducted at timepoints as specified in Table 3 and Table 4. At any scheduled timepoint, several spirometry be carried out by the patient for up to a maximum of the device will be conducted at timepoints as specified by the device will be conducted at timepoints as specified in Table 3 and Table 4. At any scheduled timepoint, several spirometry data specified in Table 3 and Table 4. At any scheduled timepoint, several spirometry efforts will be carried out by the patient for up to a maximum of 8 efforts. Of these 8 efforts, a best effort is identified by the device. The SDTM datasets will contain all efforts produced at each scheduled timepoint, with an indicator variable showing which effort was determined the best by

Generally, for all endpoint analyses of lung function data, the best effort will be used for analysis. The exception to this rule is the time to recovery exploratyory endpoint (See section 4.4.2) which will use the all efforts data to more precisely identify the time in which a patient returns to 15% of their baseline result.

## **Primary Efficacy Measure** 4.2

## Maximum fall from post-dose, pre-exercise baseline in FEV<sub>1</sub> 4.2.1

The maximum percentage fall during the 60-minute assessment period, prior to the use of rescue medication, will be calculated at Visit 3 and Visit 4. Only acceptable and borderline acceptable quality FEV1 measurements will be considered.

### **Secondary Efficacy Measures** 4.3

# Derivation of responder status in post exercise FEV<sub>1</sub> (10% threshold)

A binary response variable will be assigned to identify subjects with a maximum percentage fall in FEV<sub>1</sub> post-exercise of <10% separately at Visit 3 and Visit 4:

- Protected: Maximum percentage fall from post-dose, pre-exercise baseline in FEV<sub>1</sub> up to 60 minutes post-exercise challenge <10%
- Not Protected: Maximum percentage fall from post-dose, pre-exercise baseline in FEV<sub>1</sub> up to 60 minutes post-exercise challenge  $\geq$ 10%

The maximum percentage fall will be defined as per the primary endpoint in Section 4.2.1. If a subject has a missing maximum percentage fall from post-dose, pre-exercise baseline in FEV1

Derivation of responder status in post exercise FEV1 (20% threshold)

The secondary endpoint on responder status as detailed in section 4.3.1 will be repeated based on a 20% threshold:

• Protected: Maximum percentage fall for to 60 minutes

- Not Protected: Maximum percentage fall from post-dose, pre-exercise baseline in FEV<sub>1</sub> up to 60 minutes post-exercise challenge  $\geq$ 20%

If a subject has a missing maximum percentage fall from post-dose, pre-exercise baseline in FEV1 up to 60 minutes post-exercise challenge, then they will be classified as a nonresponder.

## 4.4.2

Time to recovery in post-exercise FEV<sub>1</sub>
covery at each of Visits 3 (period 1)
from the end time of the vithin 100 Time to recovery at each of Visits 3 (period 1) and 4 (period 2) will be derived as the time (minutes) from the end time of the exercise challenge test to the time in which the FEV<sub>1</sub> result returns to within 10% of the value recorded at the post-dose, pre-exercise baseline.

For time to recovery endpoints, the actual time will be used and will consider all efforts produced that are of an acceptable, or borderline acceptable quality. This will allow greater precision in identifying the time to recovery compared to using the best efforts for each nominal timepoint. Please see Section 4.1.10 for a summary of best effort and all effort spirometry data

If a subject has not observed a fall greater than 10% of the post-dose pre-exercise baseline in their post-exercise challenge test by 60 minutes, they will be left censored at 0 minutes. Subjects with an observed fall and have required rescue medication during the post-ECT assessments will be censored at the time of receiving rescue medication. Subjects who do not recover to within 10% of the post-dose, pre-exercise baseline will be censored at their last assessment taken at the visit.

Once the event time has been derived for each subject and period, period preferences will be assigned as follows:

Statistical Analysis Plan Avillion

| Time to event | Period preference |
|-------------------|-------------------|
| $t_1 < t_2$ | Period 1 |
| $t_1 > t_2$ | Period 2 |
| $t_1 = t_2^{[a]}$ | No preference |

 $t_i$  = time to event in period i. If a subject is censored at a particular period,  $t_i$  represents the time to censoring.

<sup>[a]</sup> If event times have required censoring and it cannot be determined which period is of preference, then *no period preference* will be assigned for that subject. A working example is as follows: If a subject required rescue medication at 10 minutes post-ECT in period 1, and at 20 minutes in period 2, then we have censored event times of [>10 minutes, >20 minutes] for  $t_1$  and  $t_2$ , respectively. Since  $t_1 - t_2$  spans a range of possible outcome, that includes a difference of 0 minutes (-10 minutes, + $\infty$  minutes), this subject is classified as having no period preference for their time to recovery.

# 4.4.3 Derivation of FEV<sub>1</sub> AUC<sub>0-30min</sub>

FEV<sub>1</sub> AUC<sub>0-30min</sub> will be derived for the changes from the post-dose, pre-exercise baseline using the trapezoidal rule and will be normalized by dividing by the actual time (in minutes) from the exercise challenge test to the last included measurement, scheduled at 30 minutes post-exercise challenge at each of Visits 3 and 4. Only FEV<sub>1</sub> results prior to the use of rescue medication will be considered when calculating FEV<sub>1</sub> AUC<sub>0-30min</sub>.

be considered when calculating FEV<sub>1</sub> AUC<sub>0-30min</sub>. 
$$AUC_{0-30 \text{ minutes}} = \frac{1}{t_N - t_0} \times \sum_{i=1}^N \frac{(y_{i-1} + y_i) \times (t_i - t_{i-1})}{2}$$

For FEV<sub>1</sub> change from baseline results  $y_i$  recorded  $t_i$  minutes after the exercise challenge test (actual clock time at i=0,1,2,...,N actual timepoints. If all post-exercise timepoints are available, then N=4, to corresponds to the end time of the exercise challenge test and  $y_0=0$ . Only FEV results of 'acceptable' or 'borderline acceptable' (investigator assigned) quality will be used in the derivation of FEV<sub>1</sub> AUC<sub>0-30 minutes</sub>. If a FEV<sub>1</sub> result is missing or recorded in the database, but assigned an 'unacceptable' quality grade at the scheduled assessment, then the assessment will be excluded from the calculation of FEV<sub>1</sub> AUC<sub>0-30 minutes</sub>. To calculate FEV<sub>1</sub> AUC<sub>0-30 minutes</sub>, there must be at least 1 non-missing post-dose FEV<sub>1</sub> within 0 to 30 minutes post-dose. Missing FEV<sub>1</sub> post-dose measures will not be imputed.

#### 4.5 Safety variables

#### 4.5.1 Vital signs

extension of such application le. The following vital signs measurements are conducted throughout the study and as per Table 3 and Table 4.

- Pulse rate (beats/min)
- Systolic blood pressure (mmHg)
- Diastolic blood pressure (mmHg)

Any clinically significant changes in vital signs are recorded as an AE if applicable.

Changes from baseline to each post-ECT timepoint in vital sign parameters will be calculated based on the period-specific baseline result (4.1.5.2) for each visit 3 and visit 4.

### Adverse events (including Serious Adverse Events 4.5.2

#### 4.5.2.1 **Definition of adverse event**

An AE is the development of any untoward medical occurrence in a subject or clinical study subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom (e.g., nausea, chest pain), or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

The term AE is used to include both serious and non-serious AEs and can include a deterioration of a pre-existing medical occurrence. An AE may occur at any time, including the screening period, even if an orandomized treatment has been administered.

#### 4.5.2.2 Definitions of serious adverse event

An SAE is an AE occurring during any study phase (i.e., after the signing of the informed consent/assent through to the safety follow-up TC), that fulfills 1 or more of the following criteria:

- Results in death
- as immediately life-threatening

Requires in-patient hospitalization or prolongation of existing hospitalization

- Results in persistent or significant disability or incapacity
- Is a congenital abnormality or birth defect
- Is an important medical event that may jeopardize the subject or may require medical intervention to prevent 1 of the outcomes listed above

All SAEs will be identified by the investigator and entered in the eCRF. The 'Serious?' field will be set to 'Y'.

## 4.5.2.3

ere
Serious

- Yes or no
Investigator causality rating against the range mixed treatment

- Yes or no
Cion taken regarding randomized treatment

Dose not changed
Drug interrupted
Drug permanently discontinue AEs and SAEs will be collected from time of signature of informed consent/assent, through the safety follow-up period.

The following variables will be collected for each AE:

- Outcome Otto
  - - Recovered/resolved with sequelae
  - Not recovered/not resolved

#### 4.5.2.4 Adverse events data handling

Adverse events will be reported as starting during screening if the AE start date is prior to the

If an AE has a missing onset date, then, unless the stop date of the AE indicates otherwise, this will be considered as treatment emergent. Similarly, if an AE has a partial onset date, then unless the partial onset date or the stop date indicates otherwise this treatment emergent. AEs will be represented to the stop date indicates otherwise this treatment emergent.

programm or stop dates at stop dates at the copy of the programm of the part o AE will be summarized under the BDA MDI treatment group.

Please refer to Section 4.1.9 for the imputation rules to programmatically determine the classification of AEs when there is partial start and/or stop dates recorded.


Statistical Analysis Plan Avillion

## 4.5.3 Laboratory Safety Variables

The following laboratory variables described in Table 5 Laboratory Safety Variables will be collected at screening and at unscheduled visits, if required:

**Table 5 Laboratory Safety Variables** 

| Hematology/Hemostasis (whole blood) | Clinical Chemistry (serum or plasma) Albumin Alanine transaminase Alkaline phosphatase Aspartate transaminase Bilirubin, total Calcium, total |
|---|---|
| Basophils (%) | Albumin |
| Basophils Abs | Alanine transaminase |
| Eosinophils (%) | Alkaline phosphatase |
| Eosinophils Abs | Aspartate transaminase |
| Hemoglobin | Bilirubin, total |
| Hematocrit | Calcium, total |
| Mean Corpuscular Hemoglobin | Chloride |
| Mean Corpuscular Hemoglobin Concentration | Cholesterol; Otal |
| Mean Corpuscular Volume | Greatinine |
| Monocytes (%) | Creatine kinase |
| Monocytes Abs | Gamma-glutamyl transpeptidase |
| Neutrophils (%) | Glucose (random) |
| Monocytes Abs Neutrophils (%) Neutrophils Abs Red blood cells (erythrocytes) White blood cells (leukocytes) Platelet count Lymphocytes Abs | Magnesium |
| Red blood cells (erythrocytes) | Phosphate |
| White blood cells (leukocytes) | Potassium |
| Platelet count | Protein, total |
| Lymphocytes Abs Lymphocytes (%) | Sodium |
| Lymphocytes (%) | Triglycerides |
| Urine | Urea |
| Urine β-hCG pregnancy (at Visit 3) <sup>a</sup> | Serum β-hCG pregnancy (Visit 1, 4 and PDV) <sup>a</sup> |
| Urine hemoglabin | |
| Urine erythrocytes | |
| Urine protein | |
| Ur ne albumin | |
| Urine glucose | |

Abbreviations: Abs=absolute;  $\beta$ -hCG= $\beta$ -human chorionic gonadotropin; PDV=premature discontinuation visit <sup>a</sup>  $\beta$ -hCG pregnancy testing for women of childbearing potential only

#### 4.5.4 12-lead electrocardiogram

A resting 12-lead ECG is performed at Visit 1 (Table 2). The 12-lead ECG is obtained using a Additionally, ECG results are collected pre-dose and post-exercise challenge at Visit 2 Visit 3 and Visit 4. The maximal heart rate is recorded during the exercise challenge test and entered on the eCRF.

Changes from baseline in mean heart rate (beats/min), pulse rate interval (msec), QRS duration (msec), QT interval (msec), QTcB interval (msec), QTcF interval (msec) and RR interval (msec) will be calculated at Visit 3 and Visit 4, using the period-specific pre-dose baseline.

#### 4.6 Other variables

#### 4.6.1 Concomitant medications

The collection and recording of all concomitant medication, including all pre-enrollment asthma therapies, are performed at the visits detailed in Table 2.

If a concomitant medication is recorded with partial start date and/or end date of administration, a conservative approach will be considered such that unless it can be unequivocally determined that the medication started and ended prior to the first dose of randomized study drug, based on available information from the partial date(s), the medication will be classified as concomitant. To facilitate this decision-making process programmatically, the imputation process defined in section 4.1.9 will be considered.

### 4.6.2 Withdrawal from study

Reasons for premature withdrawal from the study for randomized subjects are collected on the eCRF and include the following fields:

- Patient Decision
- Adverse Event
- Severe non-compliance to protocol
  - Condition under investigation worsened
- Lack of Therapeutic Response
- Development of study specific discontinuation criteria
  - A severe exacerbation event
  - Pregnancy

- Subject lost to follow-up
- Other

Patients who withdraw prior to randomization, or are lost to follow-up following Visit 4 (i.e. the safety follow-up call) will have their end of study status collected in the eCRF under the following fields:

Adverse Event
Completed
Death
Lost to Follow-Up
Protocol Deviation
Screen Failure
Withdrawal by Subject
Withdrawal by Parent/Guardian
Other (specify)

4.6.3 Screen Failures
Screen failures
Screen failures are subjects who do not failfill the eligibility criteria for the study, and therefore must not be randomized. These subjects should be recorded as a 'Screen Failure' on the disposition of the CRF page. Subjects who are agreed followed:

Randomized subjects who do not failfill the eligibility criteria for the study, and therefore must not be randomized. These subjects should be recorded as a 'Screen Failure' on the disposition of CRF page. Subjects who are agreed followed:

therefore must not be randomized. These subjects should be recorded as a 'Screen Failure' on the disposition eCRF page. Subjects who are screen failures will not be rescreened.

Where a subject does not meet all the eligibility criteria but is randomized in error, or incorrectly started on treatment, the investigator should inform the medical monitor immediately, and a discussion should occur between the medical monitor and the investigator regarding whether to continue or withdraw the subject in the study. The medical monitor must ensure all decisions are appropriately documented. All subjects randomized in error will be analyzed in accordance with the FAS and Safety analysis set definitions (Section 2).

# 4.6.4 Maximum fall from post-dose, pre-exercise baseline in FEV<sub>1</sub> at Visit 2

rose-uose, pre-exercise baseline in FEV<sub>1</sub> at Visit in Fever at Visit 2 for all subjects as per the derivation given in Section 4.2.1. The post-dose pre-exercise baseline is defined as the 30 minute post-dose measurement taken prior to exercise at Visit 2.

#### **5.** ANALYSIS METHODS

#### 5.1 **Statistical Considerations**

extension of such application All personnel involved with the analysis of the study will remain blinded until database lock and identification of protocol deviations are identified.

Analyses described within this Statistical Analysis Plan will be performed by

#### 5.1.1 **Estimands**

Two estimands are of interest in this study:

The primary estimand of interest is the Efficacy Estimand, defined as the effect of the randomized treatments in all subjects and in the absence of intercurrent events which may impact the interpretation of the treatment effect. This estimand could be considered a whileon-treatment strategy or a hypothetical strategy as defined in the draft\(\)ICH E9 Addendum. Per protocol, subjects will have serial spirometry procedures stopped prematurely if the postexercise FEV<sub>1</sub> result drops below 40% and requires rescue therapy (SABA). Rescue therapy in this scenario is not an intercurrent event since reaching the maximum fall has triggered administration of rescue. However, rescue medication use that is prior to the first spirometry reading being taken or if there are no spirometry data that meet ATS/ERS acceptability criteria prior to the use of rescue medication will constitute an intercurrent event. This estimand targets the treatment difference in a scenario where the intercurrent event does not occur, such that outcomes for subjects without the intercurrent event are as observed, and outcomes for subjects with the intercurrent event are treated as though they had completed the observation period. A while on treatment strategy will be used such that missing maximum percentage fall data will be assumed missing at random (MAR) and handled by the direct likelihood methods of the mixed effects model.

Missing data not preceded by an intercurrent event, such as subjects who withdraw from study will be assumed to be MAR under the efficacy estimand.

The efficacy estimand will be applied to the primary analyses and exploratory analyses of: Maximum percentage fall from post-dose pre-exercise FEV<sub>1</sub>, up to 60 minutes following the

prior to any post-exercise challenge spirometry measures, or have no spirometry data the meet ATS/ERS acceptability criteria prior to the use of negative outcome. In the The second estimand of interest is the attributable estimand, defined as the effect of treatment meet ATS/ERS acceptability criteria prior to the use of rescue medication will be considered a exercise FEV<sub>1</sub> will be imputed using a reference based approach as detailed in section 5.2.9.

The analysis of the primary endpoint under the attributable estimand will be considered a supportive analysis to assess robustness of conclusions made under the efficacy estimand.

of such application Additionally, the secondary and exploratory responder analyses as specified in sections 5.2.5.1 and 5.2.7.1 will be conducted under the attributable estimand. Patients with missing postexercise challenge FEV<sub>1</sub> measurements will be imputed as non-responders.

#### 5.1.2 Type I error control

Two subgroups of approximately equal size will be included in the study, 1 subgroup of subjects on SABA prn only and the other subgroup on low-dose ICS maintenance therapy according to GINA guidelines. All primary, secondary and exploratory analyses will be repeated on each of these subgroups of interest. For the primary analyses in each subgroup, a sequential testing strategy will be adopted, controlled at  $\alpha = 5\%$  for each comparison. The subgroup comparisons will be conducted in the following sequence:

- 1. Overall population (SABA prn only OR low-to-medium dose ICS plus SABA prn background therapy)
- 2. Subjects taking SABA prn only for background therapy
- 3. Subjects taking low-to-medium dose ICS plus SABA prn for background therapy

If a comparison is significant (alpha=0.05, 2-sided) testing will proceed to the next comparison. Comparisons will stop if a non-statistically significant result occurs. All comparisons are of superiority of BDAMDI 1609/180 versus Placebo MDI. Please refer to section 5.2.4 for further detail on the primary analysis.

## **Treatment groups** 5.1.3

Descriptive summaries and analyses of endpoints listed below will be grouped by treatment. As subjects will receive both BDA 160/180 MDI and Placebo MDI. Subjects will be represented by the treatment they receive at each visit. Therefore, post-randomization analyses of endpoints will not be broken down by visits, since visits will be mutually exclusive per subject and their dosed treatment combinations.

## Analysis methods 5.2

All tests will be 2-sided and conducted at 5% level of significance unless otherwise stated.

When appropriate, statistical analysis models will be adjusted to include the stratification factor of background ICS which will be used to describe the populations of clinical interest for the study. All subjects who are randomized and are part of the FAS will be analyzed according to the strata they were allocated to in IVRS/IWRS. Any subjects who are miss-stratified will be identified as important protocol deviations and listed in the CSR.

In addition to the analyses described below, all variables will be summarized descriptively where appropriate.

mule analysis (n); Mean; Standard Deviation; Median; Maximum; Maximum. Summaries of categorical endpoints will include the absolute counts and percentage, with the denominator used in the percentage calculation clearly defined in the footnote of the table. Unless stated otherwise, the denominator will be the number of subjects in the analysis set used for the descriptive summary.

5.2.1

#### 5.2.1 **Subject Disposition**

Subject disposition will be summarized for all subjects who have been enrolled and have provided informed consent. The number of subjects who were enrolled, screened and screen failed will be summarized. The number and percentage of subjects will be presented by the following categories; randomized, not randomized (and reasons), randomized who received study treatment, randomized who did not receive study treatment (and reasons), completed, and discontinued the study (and reasons). If the reason for premature discontinuation is "Development of study specific discontinuation criteria" the specify field, which contains standard text, will be reported as a sub-field in the summary table. For categories that are postrandomization, summaries will be further split by treatment sequence.

A separate table will present the number and percentage of subjects randomized to each treatment sequence, by country and center. This table will be based on the FAS.

A descriptive summary of the number subjects allocated to the safety analysis set and FAS will be presented by treatment sequence. This summary will use the all randomized subjects population.

### **Demographic and Baseline Characteristics** 5.2.2

The summary of demographic and baseline characteristics will be performed on the FAS and will be summarized by treatment sequence (including total across sequence groups).

Demographic characteristics of age (years), sex, race and ethnic group will be summarized descriptively.

Subject height (cm), weight (kg) and BMI (kg/m<sup>2</sup>) will be summarized by treatment sequence

Maximal heart rate at some (including Maximal heart rate at screening Visit 1 and Visit 2 will be summarized by treatment sequence (including total across sequence groups). At Visits 3 and 4, the maximal heart rate will be summarized descriptively by treatment group.

Lung function endpoints of pre-ECT FEV<sub>1</sub> (L), FVC (L) and FEV<sub>1</sub>/FVC (%) will be summarized at Visit 1 and Visit 2 descriptively, within treatment sequence and across treatment sequences. Additionally, maximum percentage fall in post-dose pre-exercise challenge will be presented for Visit 2 by treatment sequence and overall. All lung function data collected at screening will be listed.

Medical (past and current) and surgical histories will be summarized by MedDRA preferred term within MedDRA system organ class. The MedDRA version used for coding will be provided in the corresponding programmed output footnotes.

Smoking status will be summarized categorically as the number of subjects who have never smoked, are current smokers or are former. Nicotine pack years, e-cigarette pack years and total (nicotine + e-cigarette) pack years will be summarized as continuous empoints.

Asthma history variables collected on the eCRF will be summarized descriptively. Time since diagnosis of asthma will be summarized as a continuous scale and present the median, minimum and maximum result by treatment sequence.

## 5.2.3

Treatment exposure will be listed for all subjects.

## 5.2.4

Analysis of the primary endpoint and mum percentage fall from post-docation post-docation spost-exercise challenges fixed effects The maximum percentage fall from post-dose, pre-exercise baseline in FEV<sub>1</sub> observed up to 60 minutes post-exercise challenge will be analyzed with a mixed effect model including categorical fixed effects for treatment period and treatment sequence. Continuous covariates include period-specific pre-dose baseline FEV<sub>1</sub> and average pre-dose baseline FEV<sub>1</sub> in order to eliminate cross-level bias whilst using pre-treatment baselines (Kenward and Roger, 2009). A random subject within treatment sequence effect will be specified. Estimated treatment differences in maximum percentage fall from post-dose pre-exercise FEV1 up to 60 minutes post-ECT will be presented from the model, along with associated 95% confidence intervals (CIs) and 2-sided p-values.

The corresponding hypotheses for the primary analysis are as follows:

 $H_{01}$ : Difference between treatments = 0,

 $H_{A1}$ : Difference between treatments  $\neq 0$ .

The primary treatment comparison of BDA MDI 160/180 versus placebo MDI for the maximum percentage fall from post-dose, pre-exercise baseline in FEV<sub>1</sub> observed up to 60 minutes post-exercise challenge will be conducted on the FAS and include all data up to study withdrawal as per the Efficacy Estimand. Missing results for maximum percentage fall in

FEV<sub>1</sub> are unlikely (i.e., rescue medication will most likely occur after to the collection of the 5 minutes measure) and will be assumed to be missing at random. Based on previous studies it is highly unlikely that a subject will require rescue medication prior to their first post-ECT measurement (Ostrom et al 2015).

The primary analysis will be repeated on the subgroups of clinical interest (SABA prn alone; low-to-medium dose ICS plus SABA prn). To control the overall type-I error controlled at 5%, a hierarchical testing strategy will be adopted. The treatment comparisons of BDA MDL 160/180 versus placebo MDI will be conducted on the subject sub-populations of the FAS in the sequence given below:

- 1. Overall population (SABA prn only OR low-to-medium dose ICS plus SABA prn background therapy)
- 2. Subjects taking SABA prn only for background therapy
- 3. Subjects taking low-to-medium dose ICS plus SABA prn for background therapy

If a comparison is significant (alpha=0.05, 2-sided), testing will proceed to the next comparison. Comparisons will stop if a non-statistically significant result occurs. All comparisons are of superiority. Least squares mean estimates, 95% confidence intervals and associated p-values of the treatment difference will be calculated for the subgroups of clinical interest by additionally adjusting for background therapy and background therapy\*treatment group interaction in the mixed model.

All subjects who are randomized and are part of the FAS will be analyzed according to the ICS stratum they were allocated to in XVRS/IWRS in this primary analysis. A sensitivity analysis will be conducted based on subjects' actual strata to assess the impact of missstratification on the model results.

A forest plot will be created showing the difference in least squares mean estimates and associated 95% confidence intervals for the Overall, ICS and non-ICS subgroups.

## Analysis of the secondary efficacy variables 5.2.5

In addition to the analyses described below, all variables will be summarized descriptively said infere some estimand. The analyses in the rest (SABA prin alone; low-to-medium do applied to the secondary efficacy analyses.

5.2.5.1 Responder analyses.

The oddwhere appropriate. All descriptive and inferential analyses will be described in accordance with the attributable estimand. The analyses will be repeated in the key subgroups of clinical interest (SABA prn alone; low-to-medium dose ICS plus SABA prn). No type-I error control

## Responder analysis in post-exercise FEV<sub>1</sub>

The odds of being protected against EIB (i.e., having a maximum percentage fall in FEV<sub>1</sub> post-exercise challenge of <10%) will be analyzed using a generalized linear mixed model with logit link function to compare the treatments. The model will be adjusted with fixed

effects for treatment, treatment period and treatment sequence, period specific pre-dose baseline FEV<sub>1</sub> and average pre-dose baseline FEV<sub>1</sub> as continuous covariates, and a random

J.2.6 Analysis of safety variables

The safety analyses will include all data collected prior to study withdrawal and will use the safety analysis set. Safety data collected during screening will be listed separately.

5.2.6.1 Adverse events

Adverse events will be summarized by treatment signed to the event by the Marking ecent version. recent version available at the time of database lock. The following summaries will be included:

- Number of subjects with any AE in any category during randomized treatment period.
- Incidence of adverse events in the randomized treatment period by SOC and PT.
- Number of subjects with AE with outcome of death by SOC and PT.
- Serious adverse events during the randomized treatment period by SOC and PT.

All adverse events data collected including adverse events occurring during screening will be listed for each subject in the safety analysis set.

A separate listing will be produced detailing any other significant adverse events as identified by the scientific review prior to database lock and unblinding of the trial.

### Vital signs 5.2.6.2

Absolute values and changes from baseline in vital signs variables (Section 4.5.1) will be descriptively summarized by timepoint within treatment group. Vital signs will be listed for all subjects in the safety analysis set.

## Clinical chemistry and hematology

All laboratory data collected during the screening period and at unscheduled visits will be listed for subjects in the safety analysis set.

#### 5.2.6.4 Electrocardiogram

ECG parameters will be summarized as absolute values and changes from baseline by

wno take disallowed concomitant medications during the study, will be presented by standardized medication name, within generic class (WHO Drug dictionary text) for each treatment group.

Listings will be grouped by prior medication, medication treatment period.

Listings will be grouped by prior medication, medication occurring during the randomized treatment period.

#### 5.2.7 **Analysis of exploratory variables**

In addition to the analyses described below, all variables will be summarized descriptively where appropriate. All descriptive and inferential analyses will be described in accordance with the Efficacy Estimand, unless states otherwise in the endpoint specific subsections (below). The analyses will be repeated in the key subgroup of clinical interest (SABA prn alone; low-to-medium dose ICS plus SABA prn) No type-I error control is applied to the exploratory efficacy analyses.

# Responder analysis in post-exercise FEV<sub>1</sub> (20% threshold) 5.2.7.1

The odds of having a maximum percentage fall in FEV<sub>1</sub> post-exercise challenge of <20% will be separately analyzed using a generalized linear mixed model to compare treatments as specified in Section 5.2.5.1. Any subjects who required rescue medication prior to the 5 minute lung function assessment will be considered a non-responder, in accordance with the attributable estimand for responder analyses. This analysis will be repeated for subgroups of clinical interest by additionally adjusting for background therapy (non-ICS, ICS) and background therapy\*treatment group interaction.

Additionally, a scatter plot of maximum percentage fall from post-dose pre-exercise FEV<sub>1</sub> will be graphically represented with reference regions annotated to show the unprotected (>20% fall), partially protected (10%-20% fall) and protected (<10% fall) subjects, grouped by

Time to recovery

The median time to recovery will be reported descriptively by treatment. P-values will be calculated using Prescott's period-adjusted sign test, based on categorizing subjects period preferences (Senn 1993). Analyses will be starting of: All subjects per ICC period preferences (Senn 1993). Analyses will be stratified by background therapy categories

#### 5.2.7.3 Fall in post-exercise FEV<sub>1</sub> at individual time points

The percentage fall in FEV<sub>1</sub> post-exercise challenge will be summarized descriptively by as per the primary analysis, with an additional subject-periods will be unstructured over the time points. Only FEV<sub>1</sub> results prior to administration of rescue therapy (within the study visit) will be included in the analyses, as per the Efficacy Estimand. This analysis will be repeated for subgroups of clinical interestriction additionally adjusting for background therapy (non-ICS, ICS). hast

The mean percentage fall from post-dose pre-exercise FEV1 will be plotted at each nominal (planned) post-exercise timepoint for each treatment group. Error bars will be provided showing the mean  $\pm$  standard error.

described in Section 5.2.4 for the maximum percentage fall in FEV<sub>1</sub> without exercise pretreatment. Only the FEV<sub>1</sub> AUC<sub>0-30 min</sub> measurements prior to administration of rescue SABA therapy will be included in the analyses. This analysis will be repeated for subgroups of clinical interest by additionally adjusting for background therapy (non-ICS, ICS) and background therapy\*treatment group interaction.

### 5.2.8 Subgroup analysis

The assessment of treatment effect will also be investigated for primary and secondary endpoints in the other clinically important subgroups described in Table 6.

Table 6 Subgroup Analysis

| Group Subgroup Analysis | Subgroup |
|------------------------------------------|-------------------------------|
| Sex | Male |
| 150° | Female |
| Age group (years) | Adolescents: $\geq 12 - < 18$ |
| a la | Adults: $\ge 18 - < 65$ |
| Rivis | Elderly: >= 65 |
| BMI (kg/m²) | Median value cut-off [1] |
| Baseline FEV <sub>1</sub> | Median value cut-off [1] |

<sup>[1]</sup> Subgroup will be categorized into two groups defined by the median value observed at baseline.

For all subgroup analyses, if there are less than 10 subjects/events available within a subgroup and at least 5 subjects with data available per treatment group under comparison, or the model does not converge, then only descriptive (summary) statistics will be presented. Subgroup analyses will be further broken down into the overall population, and ICS and non-ICS key populations of interest. Subjects with insufficient data to be allocated to a subgroup category will be excluded from the subgroup analyses.

Generalized additive models (GAM) will be fit to explore any potential non-linear association between the crossover differences in the primary endpoint versus age, BMI and baseline  $EV_1$ as continuous measures. The GAM will use the gaussian link and plots will be presented showing the smoothing splines and associated 95% confidence limits.

Forest plots will be produced showing the least squares mean difference and associated 95% confidence intervals within each subgroup for the primary endpoint of maximum percentage fall from post-dose, pre-exercise baseline in FEV<sub>1</sub>.

fall from post-dose, pre-exercise baseline in FEV<sub>1</sub>.
5.2.9 Supportive analysis
5.2.9.1 Attributable estimand
Analysis under the attributable estimand will be conducted in the FAS and will act as a supportive analysis to the primary endpoint (section 5.2.4). Data that are missing will be imputed using reference-based imputation. Subjects with a missing maximum percentage fall in the 60-minute assessment period, for any visit, will be imputed using the least squares mean estimate of the maximum percentage fall in the Placebo MDI treatment group from a mixed model as specified in 5.2.4, using the observed data. The dataset of complete data, following imputation, will be re-analyzed as per section 5.2.4 and estimated treatment differences, associated 95% confidence intervals (CIs) and p-values will be provided.

### 5.2.10 **COVID-19** impacts

Tyree is an on-going treal throughout the coronavirus disease 2019 (COVID-19) outbreak. Due to the design and short study duration, it is not expected that trial data or the analyses will be greatly impacted by the pandemic. Although, it is important to be able to identify any potential intercurrent events due to COVID-19 and to be able to quantify their impact on the efficacy and safety profile of the study.

## 5.2.40.1 Missed Visits due to COVID-19

Due to the design of Tyree, a missed visit is not expected to occur. If a subject misses a Screening visit (Visit 1/1a, Visit 2/2a) then the subject has not provided suitable eligibility criteria to enroll and will not be randomized. If a subject misses Visit 3 and it is not rescheduled, then they will not have been randomized to the study and will be screen failed. If they miss Visit 4 and it is not rescheduled, then the subject will be considered as a premature withdrawal from the study and will be documented as such in the eCRF.

## 5.2.10.2 Premature discontinuation due to COVID-19

g at sion of such application ariation of extension of ex If a subject cannot continue with procedures and scheduled assessments due to COVID-19 post-randomization, they will be withdrawn from the trial and will be asked to complete the PDV. A separate listing of subjects who prematurely withdraw due to COVID-19 will be provided. The listing will detail the reason for withdrawal and relationship to COVID-19. The listing of premature withdrawals due to COVID-19 will be based on the full analysis set.

It is not expected that premature withdrawals will be related to randomized treatment. Therefore, the missing data subsequent to withdrawal will be considered as missing at random, in accordance with the efficacy estimand.

## 5.2.10.3 Assessments not done due to COVID-19 **Spirometry assessments**

Any subject that has not performed serial spirometry assessments at a post-randomization visit will be listed. The listing will provide the subject ID, the scheduled visit name and the corresponding reason for the missed assessment, detailing how COVID-19 impacted the missed assessment. The listing of missed spirometry data will be presented in the full analysis set.

Any missed spirometry data due to COVID-12 is not anticipated to be related to randomized treatment and as such, missed spirometry assessments will be considered missing at random, in accordance with the efficacy estimand.

Scheduled safety assessments

Any scheduled safety data, including clinical laboratory, pregnancy tests, ECG and vital signs that are missing due to COVID-19 will be listed for each subject. The listing will detail the safety procedure missed and its relationship to COVID-19. The listing of missed safety assessments will be presented in the safety analysis set.

## 5.2.10.4 Adverse events and serious adverse events due to COVID-19

All subjects with a suspected or confirmed diagnosis of COVID-19 will be listed. The listing with poetween an Al appropriately captured in the was serious or non-serious.

Listings of adverwill present any AEs with either a suspected or confirmed relationship to COVID-19. The relationship between an AE and COVID-19 will be determined by the investigator and appropriately captured in the eCRF. The listings will provide an indication of whether the AE

Listings of adverse events linked to COVID-19 will be based on the safety analysis set.

andomized sequence and auencies and percentages of accoving a percentage of a coving and percentages of a coving and percentages of a coving and percentages of a coving and percentages of a coving and accoving a coving a coving and accoving a coving a co

#### 6. CHANGES OF ANALYSIS FROM PROTOCOL

### **COVID-19 impacts** 6.1.1

As the TYREE protocol was finalized prior to the COVID-19 outbreak, the planned descriptive summaries as detailed in section 5.2.10 of this statistical analysis plan are not described within the protocol.

of such application It is not expected that trial data or the analyses will be greatly impacted by the pandemic and therefore no changes to the planned primary, secondary or exploratory analyses will be performed. Although, it is important to be able to identify any prospective intercurrent events Arimpa etalling the used to support any marketing authorization and the used to support and the used to support and the used to support and the used to support any marketing which may occur due to COVID-19 and be able to quantify their impact on the efficacy and safety profile of the study. As a result, patient-level listings detailing trial aspects that have been impacted due to COVID-19 will be provided, along with a high-level summary of these


atan DS. Novel albuterol multidose dry powder ed bronchoconstriction: a single-dose, double-blind, ay. Respir Med. 2015;109(11):1410-1415.

In Clinical Research. Wiley, Chichester 1993.

3. J. The use of baseline covariates in crossover studies. Biomedian of the state of the st

